CLINICAL TRIAL: NCT04573855
Title: TREATMENT WITH ANTI-SARS-COV-2 IMMUNOGLOBULIN IN PATIENTS WITH COVID-19: A PHASE I / II STUDY
Brief Title: TREATMENT WITH ANTI-SARS-COV-2 IMMUNOGLOBULIN IN PATIENTS WITH COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCL04/2020
Record Dates: First submitted 2020-09-30; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-SARS-CoV-2 immunoglobulin (Experimental): Treatment with Anti-SARS-CoV-2 immunoglobulin
  Interventions: Biological: Anti-SARS-CoV-2 immunoglobulin
- Control (No Intervention)

INTERVENTIONS:
Biological: Anti-SARS-CoV-2 immunoglobulin — Treatment with Anti-SARS-CoV-2 immunoglobulin
  Arms: Anti-SARS-CoV-2 immunoglobulin

SUMMARY:
A Phase I/II clinical trial for safety and efficacy evaluation of treatment with anti-SARS-CoV-2 equine immunoglobulin (F(ab')2) in hospitalized patients with COVID-19 not requiring of invasive ventilation support.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients diagnosed with COVID-19 by RT-PCR;
* Time between symptom onset and inclusion ≤ 10 days;
* Age ≥ 18 years and <75 years
* No indication of invasive ventilatory support at the time of randomization;
* Signature of the Informed Consent Form.

Exclusion Criteria:

* Pregnant or lactating women
* Severe comorbidity: Severe heart disease, severe COPD or O2-dependent COPD, terminal cancer.
* Any confirmed or suspected immunosuppressive or immunodeficiency state, including HIV (regardless of treatment, CD4 count or viral load status); asplenia; severe recurrent infections and chronic use (more than 14 days) of immunosuppressive medication in the last 6 months, except for topical steroids or short-term oral steroids (cycle lasting ≤14 days);
* History of anaphylaxis or severe allergic reaction;
* Previous use of any heterologous serum;
* Participation in trials of prophylactic drugs or vaccines for COVID-19;
* Administration of immunoglobulins and / or any blood products in the previous three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events related to the infusion of anti-SARS-CoV-2 immunoglobulin through CTCAE v4.0. | 28 days
Clearence of viral RNA evaluated by RT-PCR | 72 h

SECONDARY OUTCOMES:
Reduction of viral load evaluated by area under the curve of RT-PCR values | Day 0, Day 3, Day 7 and Day 14
  Viral load reduction evaluated by area under the curve of RT-PCR values
Length of hospital stay | For as long as the duration of the hospital stay
  number of days between admission and discharge
Orotracheal Intubation Rate | 28 days
  Number of patients who progressed to the use of invasive mechanical ventilation and require orotracheal intubation throughout hospitalization
Infusional reaction rate | 28 days
  number of patients who experienced adverse events after the immunoglobulin infusion
Mortality rate | 28 days
  number of deceased patients
Assessment of adverse events | 28 days
  Frequency of adverse events classified following CTCAE
Evaluation of clinical status | Day 0, Day 14, Day 21 and Day 28
  Results of a 7-point ordinal severity scale
Modulation of serum and cellular inflammatory marker | Day 0, Day 3 and Day 7.
  Exploratory analysis of the variation of inflammatory markers by ELISA/Luminex and flow cytometry, compared to baseline levels

IPD SHARING:
Plan to Share IPD: Undecided